CLINICAL TRIAL: NCT00699517
Title: A Multinational, Randomized, Double-blind Placebo Controlled Study of AVE8062 (25 mg/m2) Administered Every 3 Weeks in Patients With Advanced-stage Soft Tissue Sarcoma, Treated With Cisplatin (75 mg) After Failure of Anthracycline and Ifosfamide Chemotherapies.
Brief Title: A Study of AVE8062 in Advanced-stage Soft Tissue Sarcoma After Failure of Anthracycline and Ifosfamide Chemotherapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10145; EudraCT 2007-003592-39
Record Dates: First submitted 2008-05-07; First posted 2008-06-18 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Sarcoma
Keywords: tubulin modulator; endothelium; combretastatin; cisplatin
MeSH Terms: conditions — Sarcoma | interventions — AC 7700

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: OMBRABULIN (AVE8062)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMBRABULIN (AVE8062) — I.V. infusion followed by administration of cisplatin
  Arms: 1
Drug: Placebo — I.V. infusion followed by administration of cisplatin
  Arms: 2

SUMMARY:
The primary objective of the study is to compare the progression-free survival (PFS) in the 2 treatment arms

The secondary objectives of the study are :

* To compare the overall survival in the 2 treatment arms
* To compare the objective response rate in the 2 treatment arms
* To assess the safety profile of AVE8062 (in combination with the background cisplatin therapy)
* To assess the pharmacokinetics of AVE8062 and its main metabolite, RPR258063, using a population approach, in all patients enrolled in selected centers.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven soft tissue sarcoma
* Unresectable locoregional recurrent or metastatic soft tissue sarcoma
* Failure of a previous anthracycline-based regimen administered recommended dose and of prior ifosfamide therapy

Exclusion criteria:

* Less than 3 weeks elapsed from prior treatment with radiotherapy, surgery, or chemotherapy to the time of randomization
* Brain metastases and carcinomatous leptomeningitis
* Uncontrolled hypertension
* Known platinum hypersensitivity

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2008-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival | until event or study cut-off date (Tumor assessment every 6 weeks)

SECONDARY OUTCOMES:
Overall survival | until event or study cut-off date
Response rate | tumor assessment every 6 weeks
Safety profile | assessment every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (45):
- United States (6):
  - Investigational Site Number 840004, Santa Monica, California
  - Investigational Site Number 840003, Orlando, Florida
  - Investigational Site Number 840005, Maywood, Illinois
  - Investigational Site Number 840002, Newark, New Jersey
  - Investigational Site Number 840007, Philadelphia, Pennsylvania
  - Investigational Site Number 840001, San Antonio, Texas
- Belgium (3):
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056004, Haine-Saint-Paul
  - Investigational Site Number 056005, Liège
- Brazil (8):
  - Investigational Site Number 076007, Belo Horizonte
  - Investigational Site Number 076008, Goiânia
  - Investigational Site Number 076003, Ijuí
  - Investigational Site Number 076004, Jaú
  - Investigational Site Number 076006, Novo Hamburgo
  - Investigational Site Number 076002, Porto Alegre
  - Investigational Site Number 076005, Porto Alegre
  - Investigational Site Number 076009, Rio de Janeiro
- France (11):
  - Investigational Site Number 250008, Bordeaux
  - Investigational Site Number 250002, Dijon
  - Investigational Site Number 250004, Lille
  - Investigational Site Number 250001, Lyon
  - Investigational Site Number 250010, Marseille
  - Investigational Site Number 250006, Montpellier
  - Investigational Site Number 250007, Nice
  - Investigational Site Number 250005, Rennes
  - Investigational Site Number 250003, Saint-Cloud
  - Investigational Site Number 250009, Saint-Herblain
  - Investigational Site Number 250012, Saint-Priest-en-Jarez
- Hungary (2):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348002, Debrecen
- India (3):
  - Investigational Site Number 356005, Bangalore
  - Investigational Site Number 356003, Hyderabad
  - Investigational Site Number 356004, New Delhi
- Italy (4):
  - Investigational Site Number 380001, Aviano
  - Investigational Site Number 380003, Milan
  - Investigational Site Number 380004, Milan
  - Investigational Site Number 380002, Rozzano
- Serbia (2):
  - Investigational Site Number 891001, Belgrade
  - Investigational Site Number 891002, Kamenitz
- Spain (3):
  - Investigational Site Number 724004, Barcelona
  - Investigational Site Number 724001, Madrid
  - Investigational Site Number 724003, Pamplona
- United Kingdom (3):
  - Investigational Site Number 826001, Bebington
  - Investigational Site Number 826003, Bristol
  - Investigational Site Number 826002, Newcastle upon Tyne

REFERENCES:
- [Derived] Blay JY, Papai Z, Tolcher AW, Italiano A, Cupissol D, Lopez-Pousa A, Chawla SP, Bompas E, Babovic N, Penel N, Isambert N, Staddon AP, Saada-Bouzid E, Santoro A, Franke FA, Cohen P, Le-Guennec S, Demetri GD. Ombrabulin plus cisplatin versus placebo plus cisplatin in patients with advanced soft-tissue sarcomas after failure of anthracycline and ifosfamide chemotherapy: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 May;16(5):531-40. doi: 10.1016/S1470-2045(15)70102-6. Epub 2015 Apr 8. PMID 25864104